CLINICAL TRIAL: NCT01601964
Title: Vascular Endothelial Growth Factor Levels in Ectopic Pregnancy
Acronym: VEGF
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: BEH GynObs-1
Record Dates: First submitted 2012-05-17; First posted 2012-05-18 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Complication Following Ectopic Pregnancy
Keywords: VEGF, ectopic pregnancy.
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Follow-up or medical treatment.: medical treatment
- Surgical treatment: Surgical treatment

SUMMARY:
The aim of this study is to determine plasma Vascular Endothelial Growth Factor level and change in patient with ectopic pregnancy who needs to surgical treatment.

Patient with ectopic pregnancy diagnosed and treated with medically or surgically will be included in the study. This is an observational study.The plasma Vascular Endothelial Growth Factor level will be measured first day and two day after the diagnosis of ectopic pregnancy.

DETAILED DESCRIPTION:
This study is a prospective, observational, single-center study. Ethical approval was obtained from the Institutional Review Board. This study will be completed with 30 patients with ectopic pregnancy. An intervenous cannula will be centrifuged for 15 minutes at 1000 g within 30 minutes of collection. Aliquots of plasma will be added to eppendorf tubes and stored at -20°C.

Plasma Vascular Endothelial Growth Factor levels will be measured using a Human VEGF-A Platinum ELISA kit (bioscience company, Catalog No: 00122, Santa Clara, California, USA). All assays will be performed according to the manufacturer's instructions. The test kit sensitivity is 2.5 pg/ml. Intracycle variability is %4-6, intercycle variability is %8-10.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suspected ectopic pregnancy

Exclusion Criteria:

* hemodynamically unstable patient
* healthy pregnancy (a healthy increase in ß HCG)
* missed abortion
* incomplete abortion
* The patient who need immediate surgical treatment

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patients with ectopic pregnancy
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The primary Outcome Measure of this study is to determine plasma Vascular Endothelial Growth Factor cut-off level in patient with ectopic pregnancy who needs to surgical treatment. | 3-4 months

CONTACTS AND LOCATIONS:
Overall Officials: TANER A USTA, M.D., Principal Investigator — Bagcilar Training and Research Hospital, Istanbul, Turkey.
Locations (1):
- Bagcilar Training and Research Hospital, Istanbul, Turkey (Türkiye)